CLINICAL TRIAL: NCT01560117
Title: Multicenter Study to Evaluate the Combination of Oral Fludarabine, Mitoxantrone Und Rituximab Induction Therapy Und Rituximab Maintenance Therapy in Follicular B-Cell Lymphoma
Brief Title: Combination of Oral Fludarabine, Mitoxantrone Und Rituximab Induction Therapy and Rituximab Maintenance Therapy in Follicular B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: AGMT_NHL 9
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Follicular T-NHL Lymphoma; Rituximab Maintenance
Keywords: AGMT; NHL
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 i.v. every 2 months for 24 months

SUMMARY:
Immunotherapy with the monoclonal anti-CD20 antibody rituximab has become standard of care for patients with follicular lymphoma. However, there are still open questions regarding dosing and scheduling of rituximab, optimal type of chemotherapeutic combination partners during induction as well as the best interval and length of rituximab maintenance treatment. Fludarabine-mitoxantrone combinations have shown strong debulking activity as initial therapy followed by rituximab maintenance. While rituximab maintenance with a standard dose of 375 mg/m2 prolongs clinical remissions, administration schedules still vary: Three-monthly infusions for 2 years and two-monthly infusions for one or 2 years are most frequently used. A few pharmacokinetic data for rituximab have been reported for induction treatment. These studies have proposed a presumptive "active" level of 25.000 ng/ml in anti-lymphoma treatment. However, there is only limited information regarding maintenance treatment in patients who are in remission and have no remaining tumor load.

The aim of this trial is to investigate the effect of treatment with oral Fludarabine, Mitoxantrone und Rituximab and Rituximab maintenance on the depth of remission measured by BCL2/IgH PCR.

ELIGIBILITY:
Inclusion Criteria:

* a positive BCL2/IgH rearrangement in peripheral blood (PB) and/or bone marrow (BM)
* clinical stage III or IV, requiring treatment with one or more of the following criteria: symptoms related to the disease, hemoglobin less than 12 g/dL, platelets less than 100 G/L, progressive disease, bulky tumor of more than 10 cm

Exclusion Criteria:

* pretreatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-01; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
conversion rate of bcl-2 in blood and bone marrow defined by PCR | 3 years

SECONDARY OUTCOMES:
Number of patients with a response after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fridirk, MD, Principal Investigator — AKH Linz; Ulrich Jäger, Principal Investigator — AKH Wien

REFERENCES:
- [Derived] Jager U, Fridrik M, Zeitlinger M, Heintel D, Hopfinger G, Burgstaller S, Mannhalter C, Oberaigner W, Porpaczy E, Skrabs C, Einberger C, Drach J, Raderer M, Gaiger A, Putman M, Greil R; Arbeitsgemeinschaft Medikamentose Tumortherapie (AGMT) Investigators. Rituximab serum concentrations during immuno-chemotherapy of follicular lymphoma correlate with patient gender, bone marrow infiltration and clinical response. Haematologica. 2012 Sep;97(9):1431-8. doi: 10.3324/haematol.2011.059246. Epub 2012 Apr 17. PMID 22511498